CLINICAL TRIAL: NCT06249451
Title: SAB-Support-Study: Can Checklist-based Phone Calls Improve the Quality of Staphylococcus Aureus Bacteraemia (SAB) Management
Brief Title: Staphylococcus Aureus Bacteraemia (SAB)-Support-Study
Acronym: SABOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BB 140/23
Record Dates: First submitted 2024-01-19; First posted 2024-02-08 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Staphylococcus Aureus Bacteremia
Keywords: Staphylococcus aureus; Bacteremia
MeSH Terms: conditions — Staphylococcal Infections; Bacteremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrospective control group (n= 62) (No Intervention): Analysis of patients with the diagnosis of S. aureus-bacteraemia between 01.10.2022-01.10.2023
- Prospective quality-improvement group (n= 62) (Other): Analysis of patients with the diagnosis of S. aureus-bacteraemia between 22.01.2024-22.01.2025
  Interventions: Other: Checklist-based phone calls

INTERVENTIONS:
Other: Checklist-based phone calls — The treating doctor will be called on day 1 and 12 after SAB diagnosis to point out the standard of care (as per our evidence-based in-hospital standard operating procedure (SOP)) for SAB.
  On day 2 and 6 after SAB diagnosis, there will be additional phone calls if clinical management does not follow hospital guidelines.
  The study team will also leave comments in the medical charts of the respective patients if the management does not follow hospital guidelines.
  Arms: Prospective quality-improvement group (n= 62)

SUMMARY:
The main objective of this study is to investigate whether checklist-based close telephone consultation and process surveillance for S. aureus bacteraemia (SAB) can improve adherence to our in-house SAB-guidelines (prospective quality- improvement group).

In addition, the effects of telephone consultation on the clinical outcome of patients will be examined.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Inpatient treatment at the University Medicine Greifswald university hospital
* First diagnosis of SAB in hospital

Exclusion Criteria:

* SAB already known before admission
* Palliative management within 48 hrs after SAB diagnosis
* Death within 48 hrs after SAB diagnosis
* Hospital discharge within 48hrs after SAB diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2025-01-18 (Actual)

PRIMARY OUTCOMES:
SOP adherence, calculated as a sum score per patient with the following 8 parameters: | Hospital admission until hospital discharge (no later than day 90 after diagnosis)
  1. Drawing of follow-up blood cultures 2-3 days after start of adequate antibiotic therapy
  2. Early source control (removal of infected material or drainage of an abscess ≤ 72 hrs)
  3. Adequate search for SAB focus and metastatic manifestations
  4. TEE in patients with clinical indications (within 4 days of SAB diagnosis)
  5. Early start of specific therapy after receipt of results via phone call (≤12 hrs)
  6. Adequate dosage of antibiotic
  7. Sufficient duration of therapy (at least 14 d for uncomplicated bacteremia and 28 d for complicated bacteremia)
  8. Combination therapy with Rifampicin or Fosfomycin, when indicated

SECONDARY OUTCOMES:
Time to specific antimicrobial treatment according to guidelines concerning agent and duration | Hospital admission until hospital discharge (no later than day 90 after diagnosis)
Time to negativity of follow up blood cultures | Day of SAB diagnosis until hospital discharge (no later than day 90 after diagnosis)
Time till TEE is performed (when indicated) | Hospital admission until hospital discharge (no later than day 90 after diagnosis)
Length of hospital stay after SAB diagnosis | Day of SAB diagnosis until hospital discharge (no later than day 90 after diagnosis)
In-hospital mortality (all patients) | Hospital admission until hospital discharge (no later than day 90 after diagnosis)
In-hospital mortality (because of SAB complications) | Hospital admission until hospital discharge (no later than day 90 after diagnosis)
Hospital readmission until day 30 after SAB diagnosis (all patients) | Day of SAB diagnosis until day 30 after diagnosis
Hospital readmission until day 30 after SAB diagnosis (because of SAB complications) | Day of SAB diagnosis until day 30 after diagnosis
Hospital readmission until day 90 after SAB diagnosis (all patients) | Day of SAB diagnosis until day 90 after diagnosis
Hospital readmission until day 90 after SAB diagnosis (because of SAB complications) | Day of SAB diagnosis until day 90 after diagnosis
90-day all-cause mortality | Day of SAB diagnosis until day 90 after diagnosis
90-day mortality because of SAB complications | Day of SAB diagnosis until day 90 after diagnosis
Relapse of bacteremia until day 90 after diagnosis | Day of SAB diagnosis until day 90 after diagnosis
Quality of discharge summary (documentation and treatment plan), calculated as a sum score | Hospital admission until hospital discharge (no later than day 90 after diagnosis)
Infectious diseases consultation, when indicated (yes/no) | Hospital admission until hospital discharge (no later than day 90 after diagnosis)

CONTACTS AND LOCATIONS:
Locations (1):
- Greifswald University Medicine, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: No